CLINICAL TRIAL: NCT06532877
Title: Telephone Support Program for Patients With Advanced Gastrointestinal Cancer and Their Family Caregivers
Brief Title: Telephone Support in Advanced Gastrointestinal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern University (Other); M.D. Anderson Cancer Center (Other); Eskenazi Health (Other)
Responsible Party: Principal Investigator, Catherine Mosher, Professor of Psychology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21611; R01CA289486 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Neoplasm Malignant; Caregiver Burden
Keywords: Gastrointestinal Neoplasms; Family Caregivers; Acceptance and Commitment Therapy; Fatigue; Psychotherapy; Caregiver Burden
MeSH Terms: conditions — Gastrointestinal Neoplasms; Caregiver Burden; Fatigue | interventions — Acceptance and Commitment Therapy; Educational Status; Palliative Care

STUDY DESIGN:
Intervention Model Description: Advanced gastrointestinal cancer patient-family caregiver dyads (N = 244) will be randomly assigned in equal numbers to Acceptance and Commitment Therapy (ACT) or education/support using a stratified block randomization scheme to balance the groups by patient age (<65 vs. >=65 years) and performance status (patient-reported Eastern Cooperative Oncology Group [ECOG] scores 0 or 1 vs. 2).
Who Masked: Outcomes Assessor
Masking Description: Research staff will be blind to study condition when administering assessments to participants via phone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Across six weekly 50-minute sessions and a booster session, advanced gastrointestinal cancer patients and caregivers practice various mindfulness exercises, clarify their values, and set specific goals in alignment with their values. Through in-session and home practice of skills, participants learn new and more adaptive ways to respond to unwanted internal experiences (e.g., fatigue, distress). Participants receive handouts on session topics and a compact disc (CD) that the team developed to guide mindfulness practices.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Education/Support (Active Comparator): Across six weekly 50-minute sessions and a booster session, advanced gastrointestinal cancer patients and caregivers are directed to resources for practical and health information and contact information for psychosocial services. Sessions include an orientation to the patient's medical center and treatment team, education regarding common quality-of-life concerns experienced by cancer patients and caregivers, and an overview of medical center and community resources for addressing these concerns. The therapist also describes resources for addressing financial concerns and methods of evaluating health information available via the Internet and other modalities. Participants receive handouts summarizing session topics and are asked to review them as homework.
  Interventions: Behavioral: Education/Support

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Patients and caregivers in the acceptance and commitment therapy arm learn new and more adaptive ways to respond to difficult internal experiences (e.g., fatigue, thoughts, and feelings).
  Arms: Acceptance and Commitment Therapy
Behavioral: Education/Support — Patients and caregivers in the education/support arm discuss their cancer-related concerns and receive education on services available in their medical center and community.
  Arms: Education/Support

SUMMARY:
The goal of this clinical trial is to see if telephone support programs help patients and their family caregivers adjust to advanced gastrointestinal cancer. A new telephone counseling program that involves practicing strategies for managing stress and symptoms will be compared to a telephone program involving education on quality-of-life issues and psychosocial support. The main questions it aims to answer are:

Does our telephone counseling program lower the negative impact of patients' fatigue on their activities, emotions, and thinking abilities compared to a telephone program involving education and support? Does our telephone counseling program lower family caregivers' feelings of burden compared to a telephone program involving education and support?

Participants in both study conditions will:

Complete 6 weekly telephone sessions of counseling or education/support Complete a telephone booster session Complete 3 telephone interviews over about 5 months

DETAILED DESCRIPTION:
This trial tests the effects of telephone-delivered acceptance and commitment therapy (ACT) on patient fatigue interference with functioning and family caregiver burden in advanced gastrointestinal (GI) cancer (Aim 1) as well as secondary outcomes (Aim 2). This trial also examines increases in psychological flexibility as a hypothesized mediator of ACT's effects on patient fatigue interference and caregiver burden (Aim 3). Finally, two core aspects of psychological flexibility (i.e., mindfulness/acceptance and commitment/behavior change processes) are examined as exploratory mediators of ACT's effects on patient fatigue interference and caregiver burden (Aim 4). The investigators will recruit advanced GI cancer patients and caregivers from Indiana University Health, Eskenazi Health, MD Anderson Cancer Center, and Northwestern University hospitals. Potentially eligible patients will be mailed a study introductory letter along with a consent form. The letter will have a number to call if they do not wish to be contacted further. A research assistant will call all prospective participants who do not opt out approximately 1 to 2 weeks after the letter is mailed. The research assistant will describe the study as outlined in the consent form and answer any questions. Then the research assistant will administer an eligibility screening to those who consent to participate. With the patient's permission, the primary family caregiver will also be mailed a consent form and contacted via phone to screen for eligibility and obtain consent. Consenting patients and caregivers will complete a 35-minute individual phone assessment at baseline.

Following baseline assessments, patient-caregiver dyads (N = 244) will be randomly assigned in equal numbers to ACT or education/support using a stratified block randomization scheme to balance the groups by patient age (<65 vs. >=65 years) and performance status (patient-reported Eastern Cooperative Oncology Group [ECOG] scores 0 or 1 vs. 2). Dyads in both groups will complete six weekly 50-minute telephone sessions with the first session occurring one week after baseline. Blind interviewers will assess outcomes during 30-minute individual phone assessments at 2 weeks and 3 months post-intervention. Dyads in both conditions will also complete a 30-minute booster phone session one month after the 2-week follow-up. During the booster session, ACT therapists will reinforce and address any barriers to skill practice, and education/support therapists will review key medical center and community resources.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patient is at least 3 weeks post-diagnosis of unresectable stage III or stage IV gastrointestinal cancer (i.e., ampullary, anal, appendix, bile duct, colon, esophageal, gallbladder, liver, pancreatic, rectal, small intestine, or stomach cancer) and is receiving cancer care at one of the study sites.
* Patient is at least 18 years of age.
* Patient can speak and read English.
* Patient has an eligible, consenting family caregiver (see criteria below).
* Patient has moderate to severe fatigue interference with functioning.

Patient Exclusion Criteria:

* Patient shows significant psychiatric or cognitive impairment that would preclude providing informed consent and study participation.
* Patient reports being able to do little activity on a functional status measure.
* Patient is receiving hospice care at screening.
* Patient does not have working phone service.
* Patient has hearing impairment that precludes participation.
* Patient participated in the pilot trial testing the same intervention.

Caregiver Inclusion Criteria:

* Family caregiver identified by a gastrointestinal cancer patient who meets the eligibility criteria.
* Caregiver has significant caregiving burden.
* Caregiver lives with the patient or has visited the patient in-person at least twice a week for the past month.
* Caregiver is at least 18 years of age.
* Caregiver can speak and read English.

Caregiver Exclusion Criteria:

* Caregiver shows significant psychiatric or cognitive impairment that would preclude providing informed consent and study participation.
* Caregiver does not have working phone service.
* Caregiver has hearing impairment that precludes participation.
* Patient declines study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Fatigue Interference Subscale of Fatigue Symptom Inventory | 2 weeks and 3 months post-intervention
  Seven items are rated on 11-point scales (0=no interference to 10=extreme interference) that assess the extent to which fatigue in the past week interfered with general level of activity, ability to bathe and dress, normal work activity (including housework), ability to concentrate, relations with others, enjoyment of life, and mood. The seven items are summed with higher total scores indicating greater fatigue interference. The total score range is 0 to 70. This is the primary outcome for patients.
Short-form of Zarit Burden Interview | 2 weeks and 3 months post-intervention
  Twelve items are rated on 5-point scales (0=never to 4=nearly always) that assess personal strain and role strain due to caregiving. The 12 items are summed with higher total scores indicating greater caregiving burden. The total score range is 0 to 48. This is the primary outcome for caregivers.

SECONDARY OUTCOMES:
Patient-Reported Outcome Measurement Information System (PROMIS) Sleep-Related Impairment | 2 weeks and 3 months post-intervention
  This 8-item measure assesses the perceived interference of sleep problems with activities, mood, and cognition (e.g., difficulty concentrating or completing tasks). Each item is rated on a scale from 1 (not at all) to 5 (very much). Item #2 is reverse-scored and then the 8 items are summed with higher total scores indicating greater sleep-related impairment. The total scores are converted to T-scores with a range from 30.0 to 80.1. Higher T-scores indicate a worse outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome for patients.
PROMIS Ability to Participate in Social Roles and Activities | 2 weeks and 3 months post-intervention
  This 6-item measure assesses participants' ability to participate in social roles and activities. The items measure difficulty engaging in social and recreational activities as well as usual work (including housework). Each item is rated on a scale from 1 (never) to 5 (always) and is reverse coded. Then the six items are summed with higher total scores indicating greater ability to participate in social roles and activities. The total scores are converted to T-scores with a range from 26.7 to 65.0 with higher scores indicating a better outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome for both patients and caregivers.
PROMIS Global Health measure | 2 weeks and 3 months post-intervention
  This 10-item measure assesses participants' physical, mental, and social well-being. Items are rated on scales from 5 (excellent) to 1 (poor) and 5 (completely) to 1 (not at all). One item is rated on a scale from 5 (never) to 1 (always), and another item is rated on a scale from 5 (none) to 1 (very severe). Pain is rated on a scale from 0 (no pain) to 10 (worst pain imaginable) and recoded so that higher numbers indicate less pain. The items are then summed into Global Physical Health and Global Mental Health scores. The total scores are converted to T-scores with a range from 16.2 to 67.7 (Global Physical Health) and 21.2 to 67.6 (Global Mental Health), with higher scores indicating a better outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome for patients and caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Mosher, Ph.D., Principal Investigator — Indiana University Indianapolis
Locations (4):
- United States (4):
  - Northwestern Medicine, Chicago, Illinois
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University Health, Indianapolis, Indiana
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The dataset to be shared will include individual-level baseline, procedural-based (intervention session attendance, homework completion), and outcome data for approximately 244 patients and 244 family caregivers. Data will be collected from self-report surveys and the Electronic Medical Record (EMR). Data from scored assessments (e.g., psychosocial questionnaires) will include both raw data elements (e.g., individual item responses) and summary information (e.g., total scores) where feasible. To protect the privacy of study participants, the investigators will develop a plan for de-identification of this dataset, which will address participant identifiers, dates, variables that are administrative or sensitive in nature, unedited verbatim responses that are stored as text data, and variables with low frequencies for some values.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The research community will have access to the data no later than the time of an associated publication or end of the performance period, whichever is first.
Access Criteria: Data will be findable for the research community through the Harvard Dataverse. A data digital object identifier (DOI) generated by the Harvard Dataverse will be referenced in all publications to allow the research community easy access to the exact data used in the publication. Access to the data will be restricted to qualified researchers to prevent misuse, misinterpretation, and confusion.

REFERENCES:
- [Derived] Mosher CE, Shinn EH, Addington EL, Wu W, Bricker JB, Helft PR, Turk AA, Vater LB, Masood A, Jalal SI, Loehrer PJ Sr, Champion VL, Johns SA. Protocol of a randomized trial of acceptance and commitment therapy for patient fatigue interference and caregiver burden in advanced gastrointestinal cancer. Contemp Clin Trials. 2026 Jan;160:108168. doi: 10.1016/j.cct.2025.108168. Epub 2025 Nov 26. PMID 41314597